CLINICAL TRIAL: NCT02852213
Title: SIngle-Stage, Open-Label, Safety and Efficacy Study of Adeno-Associated Virus Encoding Human Aromatic L-Amino Acid Decarboxylase by Magnetic Resonance MR-guided Infusion Into Midbrain in Pediatric Patients With AADC Deficiency
Brief Title: A Single-Stage, Adaptive, Open-label, Dose Escalation Safety and Efficacy Study of AADC Deficiency in Pediatric Patients
Acronym: AADC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Krzysztof Bankiewicz (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Krzysztof Bankiewicz, Professor of Neurological Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0269
Record Dates: First submitted 2016-07-20; First posted 2016-08-02 (Estimated); Last update posted 2025-10-21 (Actual); Status verified 2024-08

CONDITIONS: AADC Deficiency
Keywords: AADC; gene therapy
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single treatment arm (Experimental): Single-stage dose-escalation, open-label safety study of AAV2-hAADC delivered by image-guided convection-enhanced delivery bilaterally into the substantia nigra pars compacta and the ventral tegmental area of pediatric patients with AADC deficiency. Primary aim is to determine the dose for future studies based on safety, biomarkers of pharmacological activity of AADC and clinical outcomes. Cohort 1 (3 subjects) will receive a single low dose of AAV2 hAADC. The total AAV2-hAADC dose will be infused via MR guided infusion into 4 sites in both the left and right SNc and VTA. Dose intervals will be 90 days between the first 3 subjects. Cohort 2 dose (4 subjects) will be determined by Cohort 1 results. Following Cohort 2, Cohort 3/4 will be dose and divided divided by age. Cohorts 3/4 will receive the same dose by MR guided infusion to 1-2 sites bilaterally in-between the SNc and VTA. Cohort 5 (24-47mo old) will have same vector concentration and lower volume of infusion than Cohorts 3/4
  Interventions: Drug: AAV2-hAADC

INTERVENTIONS:
Drug: AAV2-hAADC — Initially, subjects will be enrolled sequentially into 2 dose groups. 3 subjects will be enrolled in Cohort 1 and treated with a single dose of AAV2 hAADC (1.3x10 11 vg, delivered as infusate volume of up to 160μL of vector at concentration of 8.3x10 11 vg/mL) on Day 0. Enrollment in Cohort 2 may commence after the last subject in Cohort 1 is treated and followed through Month 3 post-op, with approval of the data safety monitoring board (DSMB). Cohort 2 will receive a higher dose (4.2 x 10^11 vg, 160 uL). Upon DSMB review of Cohort 1/2 results, Cohort 3 (4-12 yo) and 4 (aged >/= 13 yo) will be dosed (1.6 x 10^12 vg, 60uL) in 1-2 sites bilaterally in-between the SNc and VTA. Cohort 5 will follow (aged 24-47 months) at 1.3 x 10^12 vg, 500uL. Final safety and clinical outcome assessments will be performed 1 year post-surgery. Follow-up analysis will be performed for 2 years post-op. Subjects will be enrolled in a long-term follow-up study to assess safety and clinical status updates.
  Other Names: Adeno Virus Human Aromatic L-Amino Acid Decarboxylase

SUMMARY:
The overall objective of this study is to determine the safety and efficacy of AAV2-hAADC delivered to the substantia nigra pars compacta (SNc) and ventral tegmental area (VTA) in children with aromatic L-amino acid decarboxylase (AADC) deficiency.

DETAILED DESCRIPTION:
The Study will specifically address:

* Safety, as measured by adverse events (AEs), safety laboratory tests, brain imaging, and the relationship of AEs to study/surgical procedures or to AAV2 hAADC.
* Clinical responses to treatment with AAV2-hAADC. The primary clinical outcomes will reflect the predominant motor deficits of loss of motor function and dystonic movements.

Primary Endpoints Safety: Assessment of AE or severe AE (SAE) and its relationship to study surgery, infusion, or treatment effect (graded as definite, probable, possible, unlikely or unrelated).

* Adverse Events and Serious Adverse Events
* Post-operative MRI and/or CT (with contrast if clinically indicated)
* Clinical laboratory assessments (hematology, chemistry, immunology) Biological Activity: Demonstration of effective restoration of AADC function by assays of cerebrospinal fluid (CSF) neurotransmitter metabolites and 18-fluoro-3,4-dihydroxyphenylalanine (F-DOPA) positron emission tomography (PET) imaging.

Secondary and Exploratory Endpoints To obtain preliminary data for clinical response by assessing the magnitude and variability of changes in specific outcomes.

The principal clinical outcome measures are:

* Motor function, as assessed by the Gross Motor Function Measure (GMFM-88)
* Frequency of oculogyric episodes, as measured by a Symptom Diary

Secondary clinical outcome measures include:

• Assessment of subject disability, as assessed using the Pediatric Evaluation of Disability Inventory (PEDI); adaptive behavior, as assessed using Vineland Adaptive Behavior Scale; Patient's Global Impression of Change (PGI-C); and quality of life, as determined using the Pediatric Quality of Life Inventory (PedsQL).

Although the investigators recognize that the utility of established developmental and cognitive assessments may be limited because of the study population's severe physical disability, the investigators will use the following:

* Peabody Developmental Motor Scales 2nd edition (PDMS-2)
* Bayley Scales of Infant Development, 3rd edition.

ELIGIBILITY:
Inclusion Criteria

1. Definite diagnosis of AADC deficiency, confirmed by at least two of the following three criteria: (1) CSF neurotransmitter profile demonstrating reduced HVA and 5-HIAA, and elevated 3-OMD concentrations; (2) Plasma AADC activity less than or equal to 5 pmol/min/mL; (3) Molecular genetic confirmation of homozygous or compound heterozygous mutations in DDC.
2. Age 24 months and older.
3. Failed to derive adequate benefit from standard medical therapy (dopamine agonists, monoamine oxidase inhibitor, pyridoxine or related form of Vitamin B6), as judged by presence of residual oculugyric crises and developmental delay.
4. Documented history of motor developmental delay, with inability to walk independently without support by age 18 months.
5. Cranium sufficiently developed, with sutures closed, to enable surgical placement of SmartFrame® system on the head for MRI-guided stereotactic targeting.
6. Brain MRI does not show any conditions or malformations that are clinically significant with respect to risks for stereotactic brain surgery.
7. Parent(s)/legal guardian(s) of the subject must agree to comply with the requirements of the study, including the need for frequent and prolonged follow-up.
8. Both parents (or legal guardians) must give their consent for their child's participation in the study parents unless (i.) one parent is deceased, unknown or incompetent; (ii.) one parent is not reasonably available; or (iii.) one parent has responsibility for the care and custody of the child (if consistent with state law).
9. Baseline hematology, chemistry, and coagulation values within the normal pediatric laboratory value ranges, unless in the Investigator's judgment, the out-of-range values are not clinically significant with respect to subject's suitability for surgery.

Exclusion Criteria

1. Intracranial neoplasm or any structural brain abnormality or lesion (e.g., severe brain atrophy, white matter degenerative changes), which, in the opinion of the study investigators, would confer excessive risk and/or inadequate potential for benefit.
2. Presence of other significant medical or neurological conditions that would create an unacceptable operative or anesthetic risk (including congenital heart disease, respiratory disease with home oxygen requirement, history of serious anesthesia complications during previous elective procedures, history of cardiorespiratory arrest), liver or renal failure, malignancy, or HIV positive.
3. Previous stereotactic neurosurgery.
4. Coagulopathy, or need for ongoing anticoagulant therapy.
5. Contraindication to sedation during surgery or imaging studies (SPECT, PET or MRI).
6. Receipt of any investigational agent within 60 days prior to Baseline and during study participation.
7. Evidence of clinically active infection with adenovirus or herpes virus on physical examination.

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to surgery and gene transfer | 2 years
  Assessment of adverse events related to surgery (including intracerebral hemorrhage or stroke, CNS infection) and gene transfer (including severity of post-operative dyskinesia)
CSF neurotransmitter metabolite concentrations | 1 year
  Change in CSF neurotransmitter metabolite concentrations after gene transfer (increase in homovanillic acid (HVA) and 5-hydroxyindoleacetic acid (5-HIAA), and elevated 3-O-methyldopa (3-OMD) concentrations)

SECONDARY OUTCOMES:
Gross Motor Function Measure | 2 years
  Increase in Gross Motor Function Measure-88 (GMFM-88) score
Symptom Diary created by PI | 1 years
  Decrease in frequency and severity of oculogyric episodes
Fluorodopa PET scan | Evaluated at 3 months and 2 years
  Increase in signal in the striatum on FDOPA-PET imaging as brain AADC activity measure

CONTACTS AND LOCATIONS:
Overall Officials: Krystof Bankiewicz, MD, PhD, Study Director — OSU Professor of Neurological Surgery
Locations (3):
- United States (3):
  - University of California San Francisco, Benioff Children's Hospital, San Francisco, California
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share pertinent information with the subjects care team such that standard of care for the subject can be maintained.
Supporting Information: CSR

REFERENCES:
- [Background] Brun L, Ngu LH, Keng WT, Ch'ng GS, Choy YS, Hwu WL, Lee WT, Willemsen MA, Verbeek MM, Wassenberg T, Regal L, Orcesi S, Tonduti D, Accorsi P, Testard H, Abdenur JE, Tay S, Allen GF, Heales S, Kern I, Kato M, Burlina A, Manegold C, Hoffmann GF, Blau N. Clinical and biochemical features of aromatic L-amino acid decarboxylase deficiency. Neurology. 2010 Jul 6;75(1):64-71. doi: 10.1212/WNL.0b013e3181e620ae. Epub 2010 May 26. PMID 20505134
- [Background] Christine CW, Starr PA, Larson PS, Eberling JL, Jagust WJ, Hawkins RA, VanBrocklin HF, Wright JF, Bankiewicz KS, Aminoff MJ. Safety and tolerability of putaminal AADC gene therapy for Parkinson disease. Neurology. 2009 Nov 17;73(20):1662-9. doi: 10.1212/WNL.0b013e3181c29356. Epub 2009 Oct 14. PMID 19828868
- [Background] Fiandaca MS, Varenika V, Eberling J, McKnight T, Bringas J, Pivirotto P, Beyer J, Hadaczek P, Bowers W, Park J, Federoff H, Forsayeth J, Bankiewicz KS. Real-time MR imaging of adeno-associated viral vector delivery to the primate brain. Neuroimage. 2009 Aug;47 Suppl 2(Suppl 2):T27-35. doi: 10.1016/j.neuroimage.2008.11.012. Epub 2008 Nov 27. PMID 19095069
- [Background] Hwu WL, Muramatsu S, Tseng SH, Tzen KY, Lee NC, Chien YH, Snyder RO, Byrne BJ, Tai CH, Wu RM. Gene therapy for aromatic L-amino acid decarboxylase deficiency. Sci Transl Med. 2012 May 16;4(134):134ra61. doi: 10.1126/scitranslmed.3003640. PMID 22593174
- [Background] Caviness VS Jr, Kennedy DN, Richelme C, Rademacher J, Filipek PA. The human brain age 7-11 years: a volumetric analysis based on magnetic resonance images. Cereb Cortex. 1996 Sep-Oct;6(5):726-36. doi: 10.1093/cercor/6.5.726. PMID 8921207
- [Background] Dumas HM, Fragala-Pinkham MA. Concurrent validity and reliability of the pediatric evaluation of disability inventory-computer adaptive test mobility domain. Pediatr Phys Ther. 2012 Summer;24(2):171-6; discussion 176. doi: 10.1097/PEP.0b013e31824c94ca. PMID 22466386
- [Background] Dumas HM, Fragala-Pinkham MA, Haley SM, Ni P, Coster W, Kramer JM, Kao YC, Moed R, Ludlow LH. Computer adaptive test performance in children with and without disabilities: prospective field study of the PEDI-CAT. Disabil Rehabil. 2012;34(5):393-401. doi: 10.3109/09638288.2011.607217. Epub 2011 Oct 12. PMID 21988750
- [Background] Eapen M, Zald DH, Gatenby JC, Ding Z, Gore JC. Using high-resolution MR imaging at 7T to evaluate the anatomy of the midbrain dopaminergic system. AJNR Am J Neuroradiol. 2011 Apr;32(4):688-94. doi: 10.3174/ajnr.A2355. Epub 2010 Dec 23. PMID 21183619
- [Background] Gill SS, Patel NK, Hotton GR, O'Sullivan K, McCarter R, Bunnage M, Brooks DJ, Svendsen CN, Heywood P. Direct brain infusion of glial cell line-derived neurotrophic factor in Parkinson disease. Nat Med. 2003 May;9(5):589-95. doi: 10.1038/nm850. Epub 2003 Mar 31. PMID 12669033
- [Background] Haley, S., W. Coster, L. Ludlow, J. Haltiwanger and A. PA (1992). Pediatric Evaluation of Disability Inventory: Development, Standardization and Administration Manual. Boston, MA, Trustees of Boston University.
- [Background] Hnasko TS, Perez FA, Scouras AD, Stoll EA, Gale SD, Luquet S, Phillips PE, Kremer EJ, Palmiter RD. Cre recombinase-mediated restoration of nigrostriatal dopamine in dopamine-deficient mice reverses hypophagia and bradykinesia. Proc Natl Acad Sci U S A. 2006 Jun 6;103(23):8858-63. doi: 10.1073/pnas.0603081103. Epub 2006 May 24. PMID 16723393
- [Background] Hyland K, Clayton PT. Aromatic amino acid decarboxylase deficiency in twins. J Inherit Metab Dis. 1990;13(3):301-4. doi: 10.1007/BF01799380. No abstract available. PMID 1700191
- [Background] Hyland K, Clayton PT. Aromatic L-amino acid decarboxylase deficiency: diagnostic methodology. Clin Chem. 1992 Dec;38(12):2405-10. PMID 1281049
- [Background] Hyland K, Surtees RA, Rodeck C, Clayton PT. Aromatic L-amino acid decarboxylase deficiency: clinical features, diagnosis, and treatment of a new inborn error of neurotransmitter amine synthesis. Neurology. 1992 Oct;42(10):1980-8. doi: 10.1212/wnl.42.10.1980. PMID 1357595
- [Background] Jernigan TL, Archibald SL, Berhow MT, Sowell ER, Foster DS, Hesselink JR. Cerebral structure on MRI, Part I: Localization of age-related changes. Biol Psychiatry. 1991 Jan 1;29(1):55-67. doi: 10.1016/0006-3223(91)90210-d. PMID 2001446
- [Background] Jernigan TL, Tallal P. Late childhood changes in brain morphology observable with MRI. Dev Med Child Neurol. 1990 May;32(5):379-85. doi: 10.1111/j.1469-8749.1990.tb16956.x. PMID 2354751
- [Background] Johnston LC, Eberling J, Pivirotto P, Hadaczek P, Federoff HJ, Forsayeth J, Bankiewicz KS. Clinically relevant effects of convection-enhanced delivery of AAV2-GDNF on the dopaminergic nigrostriatal pathway in aged rhesus monkeys. Hum Gene Ther. 2009 May;20(5):497-510. doi: 10.1089/hum.2008.137. PMID 19203243
- [Background] Kells AP, Forsayeth J, Bankiewicz KS. Glial-derived neurotrophic factor gene transfer for Parkinson's disease: anterograde distribution of AAV2 vectors in the primate brain. Neurobiol Dis. 2012 Nov;48(2):228-35. doi: 10.1016/j.nbd.2011.10.004. Epub 2011 Oct 14. PMID 22019719
- [Background] Kim DS, Palmiter RD, Cummins A, Gerfen CR. Reversal of supersensitive striatal dopamine D1 receptor signaling and extracellular signal-regulated kinase activity in dopamine-deficient mice. Neuroscience. 2006;137(4):1381-8. doi: 10.1016/j.neuroscience.2005.10.054. Epub 2006 Jan 4. PMID 16388913
- [Background] Laske DW, Morrison PF, Lieberman DM, Corthesy ME, Reynolds JC, Stewart-Henney PA, Koong SS, Cummins A, Paik CH, Oldfield EH. Chronic interstitial infusion of protein to primate brain: determination of drug distribution and clearance with single-photon emission computerized tomography imaging. J Neurosurg. 1997 Oct;87(4):586-94. doi: 10.3171/jns.1997.87.4.0586. PMID 9322847
- [Background] Laske DW, Youle RJ, Oldfield EH. Tumor regression with regional distribution of the targeted toxin TF-CRM107 in patients with malignant brain tumors. Nat Med. 1997 Dec;3(12):1362-8. doi: 10.1038/nm1297-1362. PMID 9396606
- [Background] Lee HF, Tsai CR, Chi CS, Chang TM, Lee HJ. Aromatic L-amino acid decarboxylase deficiency in Taiwan. Eur J Paediatr Neurol. 2009 Mar;13(2):135-40. doi: 10.1016/j.ejpn.2008.03.008. Epub 2008 Jun 24. PMID 18567514
- [Background] Lonser RR, Schiffman R, Robison RA, Butman JA, Quezado Z, Walker ML, Morrison PF, Walbridge S, Murray GJ, Park DM, Brady RO, Oldfield EH. Image-guided, direct convective delivery of glucocerebrosidase for neuronopathic Gaucher disease. Neurology. 2007 Jan 23;68(4):254-61. doi: 10.1212/01.wnl.0000247744.10990.e6. Epub 2006 Oct 25. PMID 17065591
- [Background] Lonser RR, Walbridge S, Garmestani K, Butman JA, Walters HA, Vortmeyer AO, Morrison PF, Brechbiel MW, Oldfield EH. Successful and safe perfusion of the primate brainstem: in vivo magnetic resonance imaging of macromolecular distribution during infusion. J Neurosurg. 2002 Oct;97(4):905-13. doi: 10.3171/jns.2002.97.4.0905. PMID 12405380
- [Background] Lonser RR, Warren KE, Butman JA, Quezado Z, Robison RA, Walbridge S, Schiffman R, Merrill M, Walker ML, Park DM, Croteau D, Brady RO, Oldfield EH. Real-time image-guided direct convective perfusion of intrinsic brainstem lesions. Technical note. J Neurosurg. 2007 Jul;107(1):190-7. doi: 10.3171/JNS-07/07/0190. PMID 17639894
- [Background] Lumsden DE, Lundy C, Fairhurst C, Lin JP. Dystonia Severity Action Plan: a simple grading system for medical severity of status dystonicus and life-threatening dystonia. Dev Med Child Neurol. 2013 Jul;55(7):671-2. doi: 10.1111/dmcn.12108. Epub 2013 Mar 1. No abstract available. PMID 23448663
- [Background] Manegold C, Hoffmann GF, Degen I, Ikonomidou H, Knust A, Laass MW, Pritsch M, Wilichowski E, Horster F. Aromatic L-amino acid decarboxylase deficiency: clinical features, drug therapy and follow-up. J Inherit Metab Dis. 2009 Jun;32(3):371-80. doi: 10.1007/s10545-009-1076-1. Epub 2009 Jan 28. PMID 19172410
- [Background] Mingozzi F, Hasbrouck NC, Basner-Tschakarjan E, Edmonson SA, Hui DJ, Sabatino DE, Zhou S, Wright JF, Jiang H, Pierce GF, Arruda VR, High KA. Modulation of tolerance to the transgene product in a nonhuman primate model of AAV-mediated gene transfer to liver. Blood. 2007 Oct 1;110(7):2334-41. doi: 10.1182/blood-2007-03-080093. Epub 2007 Jul 3. PMID 17609423
- [Background] Muramatsu S, Fujimoto K, Kato S, Mizukami H, Asari S, Ikeguchi K, Kawakami T, Urabe M, Kume A, Sato T, Watanabe E, Ozawa K, Nakano I. A phase I study of aromatic L-amino acid decarboxylase gene therapy for Parkinson's disease. Mol Ther. 2010 Sep;18(9):1731-5. doi: 10.1038/mt.2010.135. Epub 2010 Jul 6. PMID 20606642
- [Background] Peden CS, Burger C, Muzyczka N, Mandel RJ. Circulating anti-wild-type adeno-associated virus type 2 (AAV2) antibodies inhibit recombinant AAV2 (rAAV2)-mediated, but not rAAV5-mediated, gene transfer in the brain. J Virol. 2004 Jun;78(12):6344-59. doi: 10.1128/JVI.78.12.6344-6359.2004. PMID 15163728
- [Background] Pfefferbaum A, Mathalon DH, Sullivan EV, Rawles JM, Zipursky RB, Lim KO. A quantitative magnetic resonance imaging study of changes in brain morphology from infancy to late adulthood. Arch Neurol. 1994 Sep;51(9):874-87. doi: 10.1001/archneur.1994.00540210046012. PMID 8080387
- [Background] Pons R, Syrengelas D, Youroukos S, Orfanou I, Dinopoulos A, Cormand B, Ormazabal A, Garzia-Cazorla A, Serrano M, Artuch R. Levodopa-induced dyskinesias in tyrosine hydroxylase deficiency. Mov Disord. 2013 Jul;28(8):1058-63. doi: 10.1002/mds.25382. Epub 2013 Feb 6. PMID 23389938
- [Background] Richardson RM, Gimenez F, Salegio EA, Su X, Bringas J, Berger MS, Bankiewicz KS. T2 imaging in monitoring of intraparenchymal real-time convection-enhanced delivery. Neurosurgery. 2011 Jul;69(1):154-63; discussion 163. doi: 10.1227/NEU.0b013e318217217e. PMID 21430597
- [Background] Richardson RM, Kells AP, Martin AJ, Larson PS, Starr PA, Piferi PG, Bates G, Tansey L, Rosenbluth KH, Bringas JR, Berger MS, Bankiewicz KS. Novel platform for MRI-guided convection-enhanced delivery of therapeutics: preclinical validation in nonhuman primate brain. Stereotact Funct Neurosurg. 2011;89(3):141-51. doi: 10.1159/000323544. Epub 2011 Apr 14. PMID 21494065
- [Background] Richardson RM, Kells AP, Rosenbluth KH, Salegio EA, Fiandaca MS, Larson PS, Starr PA, Martin AJ, Lonser RR, Federoff HJ, Forsayeth JR, Bankiewicz KS. Interventional MRI-guided putaminal delivery of AAV2-GDNF for a planned clinical trial in Parkinson's disease. Mol Ther. 2011 Jun;19(6):1048-57. doi: 10.1038/mt.2011.11. Epub 2011 Feb 22. PMID 21343917
- [Background] Russell, D. J., P. L. Rosenbaum, L. M. Avery and M. Lane (2002). The Gross Motor Function Measure (GMFM-66 & GMFM-88) User's Manual. London, Mac Keith Press.
- [Background] Salegio EA, Streeter H, Dube N, Hadaczek P, Samaranch L, Kells AP, San Sebastian W, Zhai Y, Bringas J, Xu T, Forsayeth J, Bankiewicz KS. Distribution of nanoparticles throughout the cerebral cortex of rodents and non-human primates: Implications for gene and drug therapy. Front Neuroanat. 2014 Mar 17;8:9. doi: 10.3389/fnana.2014.00009. eCollection 2014. PMID 24672434
- [Background] Sanftner LM, Suzuki BM, Doroudchi MM, Feng L, McClelland A, Forsayeth JR, Cunningham J. Striatal delivery of rAAV-hAADC to rats with preexisting immunity to AAV. Mol Ther. 2004 Mar;9(3):403-9. doi: 10.1016/j.ymthe.2003.12.005. PMID 15006607
- [Background] Su X, Kells AP, Salegio EA, Salegio EA, Richardson RM, Hadaczek P, Beyer J, Bringas J, Pivirotto P, Forsayeth J, Bankiewicz KS. Real-time MR imaging with Gadoteridol predicts distribution of transgenes after convection-enhanced delivery of AAV2 vectors. Mol Ther. 2010 Aug;18(8):1490-5. doi: 10.1038/mt.2010.114. Epub 2010 Jun 15. PMID 20551915
- [Background] Swoboda KJ, Hyland K, Goldstein DS, Kuban KC, Arnold LA, Holmes CS, Levy HL. Clinical and therapeutic observations in aromatic L-amino acid decarboxylase deficiency. Neurology. 1999 Oct 12;53(6):1205-11. doi: 10.1212/wnl.53.6.1205. PMID 10522874
- [Background] Swoboda KJ, Saul JP, McKenna CE, Speller NB, Hyland K. Aromatic L-amino acid decarboxylase deficiency: overview of clinical features and outcomes. Ann Neurol. 2003;54 Suppl 6:S49-55. doi: 10.1002/ana.10631. PMID 12891654
- [Background] Szczypka MS, Kwok K, Brot MD, Marck BT, Matsumoto AM, Donahue BA, Palmiter RD. Dopamine production in the caudate putamen restores feeding in dopamine-deficient mice. Neuron. 2001 Jun;30(3):819-28. doi: 10.1016/s0896-6273(01)00319-1. PMID 11430814
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Voges J, Reszka R, Gossmann A, Dittmar C, Richter R, Garlip G, Kracht L, Coenen HH, Sturm V, Wienhard K, Heiss WD, Jacobs AH. Imaging-guided convection-enhanced delivery and gene therapy of glioblastoma. Ann Neurol. 2003 Oct;54(4):479-87. doi: 10.1002/ana.10688. PMID 14520660
- [Background] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Background] Ziegler DA, Wonderlick JS, Ashourian P, Hansen LA, Young JC, Murphy AJ, Koppuzha CK, Growdon JH, Corkin S. Substantia nigra volume loss before basal forebrain degeneration in early Parkinson disease. JAMA Neurol. 2013 Feb;70(2):241-7. doi: 10.1001/jamaneurol.2013.597. PMID 23183921
- [Derived] Pearson TS, Gupta N, San Sebastian W, Imamura-Ching J, Viehoever A, Grijalvo-Perez A, Fay AJ, Seth N, Lundy SM, Seo Y, Pampaloni M, Hyland K, Smith E, de Oliveira Barbosa G, Heathcock JC, Minnema A, Lonser R, Elder JB, Leonard J, Larson P, Bankiewicz KS. Gene therapy for aromatic L-amino acid decarboxylase deficiency by MR-guided direct delivery of AAV2-AADC to midbrain dopaminergic neurons. Nat Commun. 2021 Jul 12;12(1):4251. doi: 10.1038/s41467-021-24524-8. PMID 34253733

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT02852213/Prot_SAP_002.pdf